CLINICAL TRIAL: NCT02137551
Title: Appointment Based Model (ABM) for Accountable Care Organization (ACO) Beneficiaries
Brief Title: ABM for ACO Beneficiaries
Acronym: ABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Pharmacists Association Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 012
Record Dates: First submitted 2014-05-02; First posted 2014-05-14 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Medication Adherence
Keywords: adherence; healthcare costs; appointment based model; accountable care organization
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABM Intervention in FQHC (Experimental): Pharmacy technicians within El Rio will implement the ABM
  Interventions: Other: ABM
- ABM Intervention in a Supermarket Pharmacy (Experimental): Pharmacists within Fry's will implement the ABM
  Interventions: Other: ABM
- Usual care (No Intervention): Patients will refill prescriptions at their usual pharmacy in the customary way.

INTERVENTIONS:
Other: ABM — The ABM involves synchronizing all medications to come due on the same say of the month and the individual receives a pre-appointment phone call from the pharmacy staff to review medications and identify any changes.
  Other Names: Appointment Based Model
  Arms: ABM Intervention in FQHC; ABM Intervention in a Supermarket Pharmacy

SUMMARY:
The primary objective of the study is to evaluate how engaging ACO beneficiaries in the appointment based model for one year impacts medication adherence and healthcare costs compared to usual care.

DETAILED DESCRIPTION:
The American Pharmacists Association (APhA) Foundation has partnered with a federally qualified health center (FQHC), a supermarket community pharmacy, and an accountable care organization (ACO) to participate in this ABM for ACO Beneficiaries initiative. The FQHC, El Rio Community Health Center pharmacy, and supermarket pharmacy, Fry's Pharmacy, will serve as implementing pharmacy study sites and will implement the ABM for beneficiaries of the ACO who utilize their pharmacies for medication refill services. The ABM involves synchronizing all medications to come due on the same day of the month and the individual receives a pre-appointment phone call from the pharmacy staff to review medications and identify any changes. The ACO will provide medical and claims data on enrolled subjects as well as a control group for the intervention population. The APhA Foundation will aggregate intervention, prescription fill, and economic data from the 3 partners in an effort to evaluate the impact of the ABM on healthcare costs and medication adherence. The APhA Foundation has an a priori intent to publish the project results.

ELIGIBILITY:
Inclusion Criteria: Individuals eligible to be enrolled in the study include those who:

* Are beneficiaries of the partnering ACO;
* Are receiving medical care at El Rio and have been since before May 1, 2013;
* Are taking 2 or more medications that are refilled on 30, 60, or 90 day schedules;
* Speak English or Spanish;
* Are at least 18 years of age; and
* Are not institutionalized (i.e., residents of nursing homes, psychiatric institutions, or prisons).

Exclusion Criteria:

* Use of a legal authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Medical costs | Baseline (for the 1 year prior to the enrollment date), During the Patient Care period (approx. 1 year following enrollment)
  Total medical costs will be collected at baseline for the year prior to enrollment and at the end of the one-year study period for the intervention year.
Pharmacy costs | Baseline (at the time of enrollment), During the Patient Care period (approx. 1 year after enrollment)
  Pharmacy costs will be collected at baseline for the year prior to enrollment and at the end of the one-year study period for the intervention year.
Medication adherence | At baseline for the one year prior to enrollment, During the 1 year patient care period
  Proportion of days covered will be calculated to determine medication adherence. Data will be collected on a quarterly basis (every 3 months beginning at enrollment).

SECONDARY OUTCOMES:
Identified Medication Related Problems | During the Patient Care period (1 year from enrollment)
  Information regarding the type of medication related problem identified at each intervention point will be reported to the sponsor on a quarterly basis and during the Patient Care period.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Kunkle, PharmD, Principal Investigator — APhA; Benjamin Bluml, BPharm, Study Director — APhA Foundation
Locations (2):
- United States (2):
  - Fry's Pharmacy Care Center, Phoenix, Arizona
  - El Rio Community Health Center, Tucson, Arizona